CLINICAL TRIAL: NCT01406405
Title: Prospective Randomized Clinical Trial Comparing PEEK and Allograft Spacers in Patients Undergoing Spinal Intervertebral Fusion Surgeries
Brief Title: PEEK and Allograft Spacers Evaluation in Spinal Fusion Surgeries
Acronym: PEEK
Status: Completed | Type: Observational
Sponsor: Justin Parker Neurological Institute (Other)
Responsible Party: Sponsor
Other Study IDs: JPNI2001-2
Record Dates: First submitted 2011-07-27; First posted 2011-08-01 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Degenerative Disc Disease
Keywords: Degenerative disc disease; spinal stenosis; herniated disc
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Intervertebral Disc Displacement | interventions — Gene Fusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PEEK cages: Patients will have fusion surgery performed using polyetheretherketone (PEEK) cages
  Interventions: Procedure: Posterior/Transforaminal Lumbar Interbody Fusion (P/TLIF), Anterior Cervical Discectomy and Fusion (ACDF)
- Allograft spacers: Patients will have fusion surgery performed using allograft spacers
  Interventions: Procedure: Posterior/Transforaminal Lumbar Interbody Fusion (P/TLIF), Anterior Cervical Discectomy and Fusion (ACDF)

INTERVENTIONS:
Procedure: Posterior/Transforaminal Lumbar Interbody Fusion (P/TLIF), Anterior Cervical Discectomy and Fusion (ACDF) — Lumbar or cervical fusion

SUMMARY:
Purpose The primary purpose of this study is to prospectively compare clinical and radiographic clinical outcomes in patients undergoing cervical or lumbar interbody fusions and randomized to receive either polyetheretherketone (PEEK) or cortical allografts.

DETAILED DESCRIPTION:
Following surgery study subjects will be evaluated at the following intervals: 3 (+/- 2 weeks), 6 (+/- 1 month), 12 (+/- 2 months), 24 (+/- 2 months) months.

ELIGIBILITY:
Lumbar Fusion Patient Group

Inclusion Criteria:

* Skeletally mature adults between 18 and 70 years old
* Patients with back and leg pain due to degenerative disc disease, scheduled for TLIF/PLIF approach utilizing an interbody spacer and supplemental posterior fixation at 1, 2 or 3 adjacent levels
* Unresponsive to conservative care over a period of at least 6 months or has progressive neurological signs and/or symptoms of neurological compromise that mandate urgent surgical intervention
* Willing and able to comply with the requirements of the protocol including followup requirements
* Willing and able to sign a study specific informed consent.

Exclusion Criteria:

* More than 3 intervertebral levels to be fused
* Posterior fixation used at more than 1 level for 1-level intervertebral fusion
* Posterior fixation used at more than 2 levels for 2-level intervertebral fusion
* Posterior fixation used at more than 3 levels for 3-level intervertebral fusion
* Any additional approaches, e.g. anterior, XLIF
* Active local or systemic infection
* Prior interbody fusion surgery at the index level
* Prior fusion at the adjacent levels
* Previous known allergy to polyetheretherketone (PEEK) or titanium alloy

Cervical Fusion Patient Group

Inclusion Criteria:

* Skeletally mature adults between 18 and 70 years old
* Patients with neck and/or arm pain due to degenerative disc disease, scheduled for ACDF approach utilizing an interbody spacer and anterior cervical plate at 1, 2 or 3 adjacent levels
* Completed at least 6 weeks of conservative therapy or has progressive neurological signs and/or symptoms of neurological compromise that mandate urgent surgical intervention
* Willing and able to comply with the requirements of the protocol including followup requirements
* Willing and able to sign a study specific informed consent

Exclusion Criteria:

* More than 3 vertebral levels to be fused
* Any additional approaches, e.g. posterior cervical fusion
* Active local or systemic infection
* Prior interbody fusion surgery at the index level
* Prior fusion at the adjacent level
* Previous known allergy to polyetheretherketone (PEEK) or titanium alloy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Boulder Neurosurgical Associates patients
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Scores | 24 (+/- 2) months
  Improvement in the Neck/Arm or Low Back/Leg Visual Analog pain Scale (VAS) scores. A 30% reduction in pain intensity will be considered to be a successful response to treatment.

SECONDARY OUTCOMES:
Clinical and Radiographic Outcomes | 3 (+/-2) weeks and 24 (+/- 2) months
  * Assessment of Neck or Lower Back Disability Scores
  * Assessment of SF-36 Health Survey
  * Assessment of restoration of vertebral height, sagittal alignment, and graft subsidence
  * Assessment of fusion rates

CONTACTS AND LOCATIONS:
Overall Officials: Alan T Villavicencio, MD, Principal Investigator — Boulder Neurosurgical Associates
Locations (1):
- Boulder Neurosurgical Associates, Boulder, Colorado, United States

REFERENCES:
- [Derived] Villavicencio AT, Nelson EL, Kantha V, Burneikiene S. Prediction based on preoperative opioid use of clinical outcomes after transforaminal lumbar interbody fusions. J Neurosurg Spine. 2017 Feb;26(2):144-149. doi: 10.3171/2016.7.SPINE16284. Epub 2016 Sep 30. PMID 27689425